CLINICAL TRIAL: NCT03786133
Title: The Subgingival Microbiota in Chronic Periodontitis Patients Affected by Type 2 Diabetes Mellitus: a Retrospective Comparative Study
Brief Title: Chronic Periodontitis Microbiota in Type 2 Diabetes Mellitus Patients
Status: Completed | Type: Observational
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Marco Montevecchi, Aggregate Professor of Periodontology, University of Bologna
Other Study IDs: periopathogensdiabetes
Record Dates: First submitted 2018-12-14; First posted 2018-12-24 (Actual); Last update posted 2018-12-24 (Actual); Status verified 2018-12

CONDITIONS: Chronic Periodontitis; Type 2 Diabetes Mellitus
Keywords: Subgingival analysis; Real-time PCR; Comparative study; Chronic Periodontitis; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Chronic Periodontitis; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- type 2 diabetics: Analysis of microbiological tests in chronic periodontitis patients with type 2 diabetes mellitus
  Interventions: Diagnostic Test: Analysis of microbiological tests
- non-diabetics: Analysis of microbiological tests in chronic periodontitis patients without type 2 diabetes mellitus
  Interventions: Diagnostic Test: Analysis of microbiological tests

INTERVENTIONS:
Diagnostic Test: Analysis of microbiological tests — Collection and comparison of microbiological data

SUMMARY:
This study is a retrospective comparative evaluation of six main periodontal pathogens and total bacterial load in chronic periodontitis patients affected or not by type 2 diabetes mellitus by polymerase chain reaction analysis.

DETAILED DESCRIPTION:
The aim of this study was to compare prevalence and bacterial load of six main periodontal pathogens among chronic periodontitis patients with and without type 2 diabetes mellitus. Porphyromonas gingivalis and Aggregatibacter actinomycetemcomitans genotypes were also investigated.

The recruitment for the study sample was performed analysing the medical records of adult patients with chronic periodontitis visited between 2010 and 2016. Eligible patients were subdivided in two balanced groups on the basis of the presence or absence of type 2 diabetes mellitus at the time of the microbiological test.

For each subject, the following data have been collected: age, gender, smoking habits, type of metabolic control of diabetes, duration of diabetes, number of missing teeth.

For each subject, four periodontal sites were studied. Probing pocket depth, sites with bleeding on probing, sites with suppuration and microbiological data were evaluated.

An individual matching on the basis of severity and extension of periodontitis was performed by pairing a diabetic patient with another non-diabetic one with the same degree of severity and extension of the periodontal disease.

Microbiological data of subgingival biofilm were analysed and compared for the examined pathogens: Aggregatibacter actinomycetemcomitans, Porphyromonas gingivalis, Prevotella intermedia, Treponema denticola, Fusobacterium nucleatum, Tannerella forsythia.

Differences in genotypes of Porphyromonas gingivalis and Aggregatibacter actinomycetemcomitans among diabetic and non-diabetic patients were also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of chronic periodontitis
* diagnosis of type 2 diabetes mellitus (only in the test group)
* the presence of at least 12 teeth (except for the third molar)
* belonging to caucasian ethnic group
* age greater than 18 years.

Exclusion Criteria:

* pregnant or lactating
* history of systemic antibiotics within 3 months prior to the microbiological testing or anti-inflammatory therapy in the month before the visit
* if they were suffering from any other systemic disease except diabetes mellitus (arthritis, ulcerative colitis, Crohn's disease, osteoporosis or osteopenia, HIV infection, hematologic diseases, neoplastic diseases, cardiovascular diseases or pathologies that could potentially interfere with the periodontitis and/or with diabetes)
* mental disorders
* if they had received periodontal treatment in the 6 months before the microbiological test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The recruitment for the study sample was performed analysing the medical records of adult patients with chronic periodontitis visited between 2010 and 2016. Eligible patients were subdivided in two balanced groups on the basis of the presence or absence of type 2 diabetes mellitus at the time of the microbiological test.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-06-10 (Actual); Primary Completion 2016-07-26 (Actual); Study Completion 2016-11-16 (Actual)

PRIMARY OUTCOMES:
Bacterial load of six main periodontal pathogens | November 16th 2016
  Bacterial load mean of six main periodontal pathogens expressed as number after a polymerase chain reaction count
Prevalence of six main periodontal pathogens | November 16th 2016
  Number of sites presenting a specific pathogen
Relative bacterial load of six main periodontal pathogens | November 16th 2016
  A mean percentage that derives from the comparison of the bacterial load to the total bacterial load
Total bacterial load | November 16th 2016
  A mean of all bacteria present in a periodontal site expressed as number after a polymerase chain reaction count

SECONDARY OUTCOMES:
Genotypes of Porphyromonas gingivalis and Aggregatibacter actinomycetemcomitans | November 16th 2016
  Genotypes of Porphyromonas gingivalis and Aggregatibacter actinomycetemcomitans were compared

CONTACTS AND LOCATIONS:
Overall Officials: Marco Montevecchi, DDS, Study Chair — University of Bologna
Locations (1):
- Alma Mater Studiorum - University of Bologna, Department of Biomedical and Neuromotor Sciences, School of Dentistry - Division of Periodontology and Implantology., Bologna, Italy

IPD SHARING:
Plan to Share IPD: Yes
Data will be available when the research will be published
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available when the research will be published
Access Criteria: On request to the main investigator

REFERENCES:
- [Derived] Montevecchi M, Valeriani L, Gatto MR, D'Alessandro G, Piana G. Subgingival pathogens in chronic periodontitis patients affected by type 2 diabetes mellitus: a retrospective case-control study. J Periodontal Implant Sci. 2021 Dec;51(6):409-421. doi: 10.5051/jpis.2100180009. PMID 34965620